CLINICAL TRIAL: NCT01428661
Title: MAGELLAN: A Multicenter, Randomized, Double-Masked, Placebo-Controlled, Parallel Study to Investigate the Safety and Efficacy of 20 Mg Tasimelteon Versus Placebo in Adult Subjects With Major Depressive Disorder Followed by a 52-Week Open-Label Extension
Brief Title: Melatonin Agonist Effects of Tasimelteon Versus Placebo in Patients With Major Depressive Disorder
Acronym: MAGELLAN
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Vanda Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VP-VEC-162-2301
Record Dates: First submitted 2011-08-31; First posted 2011-09-05 (Estimated); Results first posted 2015-06-19 (Estimated); Last update posted 2015-06-19 (Estimated); Status verified 2015-06

CONDITIONS: Major Depressive Disorder
Keywords: tasimelteon; Major Depressive Disorder; MDD; depression
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — tasimelteon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- tasimelteon (Experimental)
  Interventions: Drug: tasimelteon
- placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: tasimelteon — 20 mg once daily
  Arms: tasimelteon
Drug: placebo — once daily
  Arms: placebo

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of an 8-week double-masked treatment of tasimelteon or placebo in male and female subjects with Major Depressive Disorder.

DETAILED DESCRIPTION:
This is a randomized, parallel, double-masked, placebo-controlled, multicenter outpatient study comparing tasimelteon with placebo in the treatment of subjects with Major Depressive Disorder (MDD).

The study has three phases: the pre-randomization phase, the randomization phase, and an open-label extension phase. The pre-randomization phase comprises a screening visit where subject's initial eligibility will be evaluated. The randomization phase is comprised of an 8-week double-masked segment. Subjects meeting all entry criteria for the study will enter the randomization phase. During this phase, subjects will be asked to take either 20 mg tasimelteon or placebo for 8 weeks in a double-masked fashion. At the end of the 8-week double-masked phase, those subjects who completed the 8-week treatment phase will be offered to enroll into a 52-week open-label extension where each subject will receive daily doses of 20 mg tasimelteon.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with diagnosis of MDD, single or recurrent episode, according to DSM-IV TR criteria;
* Current episode ≥4 weeks and ≤1 year;
* CGI-Severity score ≥4 at screening and baseline.

Exclusion Criteria:

* Lifetime history of bipolar disorder (I or II), schizophrenia, schizoaffective disorder, eating disorder, or obsessive-compulsive disorder;
* Any other current Axis I (except general anxiety disorder as long as it is not considered the primary disorder) or Axis II disorder;
* A positive test for drugs of abuse at the screening visit and/or history of drug or alcohol abuse/dependence as defined in DSM-IV TR, Diagnostic Criteria for Drug and Alcohol Abuse and Dependence, within the past 12 months;
* Formal psychotherapy within 3 months of the screening visit. General supportive psychotherapy is acceptable;
* Participation in a previous tasimelteon trial. Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 507 (Actual)
Dates: Start 2011-09; Primary Completion 2013-01 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (39):
- United States (39):
  - Vanda Investigational Site, Garden Grove, California
  - Vanda Investigational Site, Irvine, California
  - Vanda Investigational Site, Los Alamitos, California
  - Vanda Investigational Site, Oakland, California
  - Vanda Investigational Site, Oceanside, California
  - Vanda Investigational Site, San Diego, California
  - Vanda Investigational Site, Sherman Oaks, California
  - Vanda Investigational Site, Torrance, California
  - Vanda Investigational Site, Denver, Colorado
  - Vanda Investigational Site, Bradenton, Florida
  - Vanda Investigational Site, Jacksonville, Florida
  - Vanda Investigational Site, Maitland, Florida
  - Vanda Investigational Site, North Miami, Florida
  - Vanda Investigational Site, Orlando, Florida
  - Vanda Investigational Site, Atlanta, Georgia
  - Vanda Investigational Site, Chicago, Illinois
  - Vanda Investigational Site, Joliet, Illinois
  - Vanda Investigational Site, Prairie Village, Kansas
  - Vanda Investigational Site, Baltimore, Maryland
  - Vanda Investigational Site, Boston, Massachusetts
  - Vanda Investigational Site, Omaha, Nebraska
  - Vanda Investigational Site, Las Vegas, Nevada
  - Vanda Investigational Site, Toms River, New Jersey
  - Vanda Investigational Site, Willingboro, New Jersey
  - Vanda Investigational Site, Brooklyn, New York
  - Vanda Investigational Site, Mount Kisco, New York
  - Vanda Investigational Site, New York, New York
  - Vanda Investigational Site, Rochester, New York
  - Vanda Investigational Site, Staten Island, New York
  - Vanda Investigational Site, Cincinnati, Ohio
  - Vanda Investigational Site, Dayton, Ohio
  - Vanda Investigational Site, Portland, Oregon
  - Vanda Investigational Site, Lincoln, Rhode Island
  - Vanda Investigational Site, Memphis, Tennessee
  - Vanda Investigational Site, Austin, Texas
  - Vanda Investigational Site, Dallas, Texas
  - Vanda Investigational Site, Salt Lake City, Utah
  - Vanda Investigational Site, Seattle, Washington
  - Vanda Investigational Site, Brown Deer, Wisconsin

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: *Tasi: subject left country (1); Placebo: sponsor request (1), subject moved (1), IMP schedule (1), subject incarcerated (1), withdrawn after receipt of medical records (1), visit schedule (1)
  **Tasi: surgery (1), visit schedule (3), +UDS (2), IMP schdule (2), prohibited meds (1), withdrew consent (1), sponsor terminated trial (175)
Groups:
- Tasimelteon: 20 mg tasimelteon capsules, PO daily for 8 weeks
- Placebo: Placebo capsules, PO daily for 8 weeks
- Open Label Tasimelteon: 20 mg capsules, PO daily for 52 weeks
Period: Double-Masked Phase
Arm/Group | Tasimelteon | Placebo | Open Label Tasimelteon
Started | 254 | 253 | 0 (Does not apply.)
Completed | 197 | 204 | 0 (Does not apply.)
Not Completed | 57 | 49 | 0
Not completed — Protocol Violation | 9 | 4 | 0
Not completed — Adverse Event | 13 | 4 | 0
Not completed — Lost to Follow-up | 14 | 14 | 0
Not completed — Withdrawal by Subject | 18 | 20 | 0
Not completed — Lack of Efficacy | 2 | 1 | 0
Not completed — *Various | 1 | 6 | 0
Period: Open Label Extension
Arm/Group | Tasimelteon | Placebo | Open Label Tasimelteon
Started | 0 (Does not apply.) | 0 (Does not apply.) | 339
Completed | 0 (Does not apply.) | 0 (Does not apply.) | 19
Not Completed | 0 | 0 | 320
Not completed — Protocol Violation | 0 | 0 | 9
Not completed — Adverse Event | 0 | 0 | 15
Not completed — Lost to Follow-up | 0 | 0 | 38
Not completed — Withdrawal by Subject | 0 | 0 | 49
Not completed — Lack of Efficacy | 0 | 0 | 24
Not completed — **Various | 0 | 0 | 185

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tasimelteon | Placebo | Open Label Tasimelteon | Total
Number analyzed (Participants) | 254 | 253 | 339 | 846
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.7 (12.61) | 42.0 (12.46) | NA (NA) — The 2 phases of the trial are being separated out so the additive total is correct for each phase. | 42.9 (12.54)
Age, Continuous [Mean (Standard Deviation); unit: years] | NA (NA) — The 2 phases of the trial are being separated out so the additive total is correct for each phase. | NA (NA) — The 2 phases of the trial are being separated out so the additive total is correct for each phase. | 44.1 (12.19) | 44.1 (12.19)
Gender [Number; unit: participants]
  Female | 161 | 171 | 0 | 332
  Male | 93 | 82 | 0 | 175
Gender [Number; unit: participants]
  Female | 0 | 0 | 222 | 222
  Male | 0 | 0 | 117 | 117

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Endpoint at Week 8 Using the Total Score of the Hamilton Depression Rating Scale (HAM-D)
Description: Hamilton Rating Scale for Depression (HAM-D) assesses the range of symptoms that are most frequently observed in subjects with major depressive disorder (MDD) on a scale from 0 to 52. Higher HAM-D scores indicate more severe levels of depressive symptoms, thus, a negative change from baseline indicates a reduction (or improvement) in depressive symptoms.
Time Frame: 8 weeks
Population: The Intent-to-Treat (ITT) Population included any subject randomized into the study that receives a dose of study medication and that has completed at least one post-baseline efficacy measurement while on study medication.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Tasimelteon | Placebo | Open Label Tasimelteon
Number analyzed (Participants) | 249 | 243 | 339
units on a scale | -8.19 (0.45) | -7.83 (0.45) | -13.6 (0.34)

ADVERSE EVENTS:
Description: One subject randomized to placebo did not take any study drug.
Arm/Group | Tasimelteon | Placebo | Open Label Tasimelteon
Serious Adverse Events (participants affected / at risk) | 2/254 | 3/252 | 6/339
Other Adverse Events (participants affected / at risk) | 38/254 | 53/252 | 74/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (N=254) | Placebo (N=252) | Open Label Tasimelteon (N=339)
Non-Cardiac Chest Pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Blood Pressure Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Staphylococcal Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis A (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cervical Vertebral Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tasimelteon (N=254) | Placebo (N=252) | Open Label Tasimelteon (N=339)
Diarrhoea (Gastrointestinal disorders) | 15 (17) | 13 (15) | 8 (12)
Dry Mouth (Gastrointestinal disorders) | 14 (15) | 10 (10) | 7 (8)
Upper Respitory Tract Infection (Infections and infestations) | 9 (9) | 15 (17) | 22 (29)
Headache (Nervous system disorders) | 29 (37) | 24 (31) | 34 (47)
Somnolence (Nervous system disorders) | 17 (19) | 16 (19) | 10 (12)
Nasopharyngitis (Infections and infestations) | 9 (9) | 12 (12) | 27 (37)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No